CLINICAL TRIAL: NCT00134537
Title: Wallis Mechanical Normalization System for Low Back Pain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zimmer Spine (Industry)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SN002-001-05
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-10

CONDITIONS: Low Back Pain
Keywords: Degenerative Disc Disease of the lumbar spine
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Interspinous process and dynamic stabilization
  Interventions: Device: Interspinous process and dynamic stabilization
- 2 (Active Comparator): Conservative Care
  Interventions: Device: Conservative Care

INTERVENTIONS:
Device: Interspinous process and dynamic stabilization — Interspinous process and dynamic stabilization
  Arms: 1
Device: Conservative Care — Medication, exercise and spinal injections
  Arms: 2

SUMMARY:
The purpose of this study is to compare improvement in low back pain with Wallis (interspinous process implant) to exercise and injections.

ELIGIBILITY:
Subjects must meet all inclusion and exclusion criteria listed below for participation in the study.

Inclusion Criteria:

* Ages 18-60; male/female.
* Diagnosis of mild to moderate degenerative disc disease (DDD), which requires:

  * back pain of at least 30/100 as measured on a visual analog scale, with or without leg (radicular) pain; and
  * radiographic confirmation of the following, as determined by computed tomography (CT), magnetic resonance imaging (MRI), discography, plain film, myelography and/or flexion/extension films: up to Modic I changes on MRI, with decreased disc height up to 50% of adjacent level, and no significant osteophytes; with or without a contained disc herniation.
* Candidate for either surgery with Wallis or aggressive conservative management.
* Requires treatment at one or two lumbar levels between L1 and L5.
* Experienced symptoms for at least three months without significant resolution.
* Has undergone a regimen of at least four weeks of anti-inflammatory medication for the current episode of back pain and had exposure to physical therapy.
* Minimum baseline Oswestry score of 30% (15/50).
* Physically and mentally able to comply with the protocol, including ability to read and complete required forms, and willing and able to adhere to the follow-up requirements of the protocol.
* Voluntarily signs the subject informed consent.

Exclusion Criteria:

* Significant neuroforaminal compression requiring discectomy or foraminotomy
* Radiographic evidence of DDD at L5-S1
* Radiographic confirmation of severe facet joint disease or degeneration.
* History of any lumbar disc treatment intended to remove the disc, e.g. surgery, intradiscal electrothermal therapy (IDET), laser or enzymes such as chymopapain.
* Clinically compromised vertebral bodies at the affected level due to current or past trauma, e.g., sustained pathological fracture or multiple fractures of vertebrae.
* Unwilling to comply with 8 weeks of physical therapy.
* Subject refuses to consider epidural or facet injections for leg or back pain.
* Active systemic infection or infection at the operative site
* Osteoporosis. The Simple Calculated Osteoporosis Risk Estimation (SCORE) questionnaire will be used to screen subjects for osteoporosis; subjects whose screening suggests risk will undergo a dual-energy x-ray absorptiometry (DEXA) scan. Subjects will be excluded if the DEXA scan results indicate a T-score equal to or worse than -2.5, in accordance with the World Health Organization definition of osteoporosis.
* Paget's disease, osteomalacia, or any other metabolic bone disease other than osteoporosis, which is addressed above
* Rheumatoid arthritis, lupus, or other autoimmune disease
* AIDS, HIV, or Hepatitis
* Known allergy to titanium, polyetheretherketone, or polyester
* Current pathological lesions, such as tumor
* Congenital lumbar spinal stenosis
* Clinically relevant instability on flexion-extension as determined by the investigator by overlaying films.
* Cauda equina syndrome
* Pregnant at time of enrollment or with plans to become pregnant within the next three years
* Concomitant conditions requiring steroid treatment or prior steroid usage for more than one of the preceding three months
* Diabetes mellitus requiring daily insulin management
* Extreme obesity, as defined by National Institutes of Health (NIH) Clinical Guidelines (body mass index [BMI] > 35)
* Fusion previously performed at the same or an adjacent level; or other instrumented spinal surgery at the operative level.
* Prior participation in study of any experimental spinal implant or treatment
* Pending litigation against a health care professional
* Life expectancy of less than three years
* History of any invasive malignancy (except for non-melanoma skin cancer), unless treated with curative intent and with no clinical signs or symptoms of the malignancy for at least 5 years
* Current or recent history of substance abuse (alcoholism and/or narcotic addiction) requiring intervention
* Spondylolysis
* Translation greater than 2 mm at the symptomatic level
* Significant scoliosis (Cobb angle > 25 degrees) or scoliosis otherwise requiring surgical correction
* Kyphosis requiring surgical correction

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2004-11; Primary Completion 2011-04 (Actual); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
To provide a safety cohort for the Prospective, Multi-center, Randomized, Active-Controlled Study of the Wallis System for the Treatment of Mild to Moderate Degenerative Disc Disease of the Lumbar Spine | 24 months

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Spine Specialists of Arizona, Phoenix, Arizona
  - Arizona Institute for Minimally Invasive Spine Care, Phoenix, Arizona
  - Spine Source, Beverly Hills, California
  - UCLA Spine Center, Santa Monica, California
  - Boulder Neurosurgical Associates, Boulder, Colorado
  - The Spine Education & Research Institute, Thornton, Colorado
  - Emory University Medical Center, Atlanta, Georgia
  - Illinois Bone & Joint Institute, Morton Grove, Illinois
  - Fort Wayne Orthopedics, Fort Wayne, Indiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Orthopaedic Associates, Towson, Maryland
  - The Orthopedic Center of St. Louis, Chesterfield, Missouri
  - Orthopedic Spine Care of Long Island, Melville, New York
  - Orthopedic Spine Associates, Eugene, Oregon
  - The Orthopedic Specialty Center (Abington Hospital), Willow Grove, Pennsylvania
  - Central Texas Spine Institute, Austin, Texas
  - TBI/ Plano Presbyterian Hospital, Plano, Texas